CLINICAL TRIAL: NCT04755556
Title: Effectiveness of Routine Physical Therapy With or Without Home Based Intensive Bimanual Training on Clinical Outcomes in Cerebral Palsy Children: A Randomized Controlled Trial
Brief Title: Effectiveness of Routine Physical Therapy With Intensive Bimanual Training in Cerebral Palsy Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-UOL-FAHS/718-XI/2020
Record Dates: First submitted 2021-02-10; First posted 2021-02-16 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; Bimanual Training
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Home Based Intensive Bimanual training
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Other): Intensive bimanual training with routine physical therapy
  Interventions: Other: home based intensive bimanual training
- control group (Other): routine physical therapy
  Interventions: Other: Routine Physical Therapy

INTERVENTIONS:
Other: home based intensive bimanual training — Home Based Intensive Bimanual Training with Routine Physical Therapy bimanual training includes. functional activities play with ball, make a dough, make beads, make blocks .Routine Physical Therapy includes stretching spastic muscles, EMS, normalizing muscle tone.
  Arms: Experimental group
Other: Routine Physical Therapy — Routine physical Therapy includes stretching spastic muscles, EMS, normalizing muscle tone.
  Arms: control group

SUMMARY:
Effectiveness of Routine Physical Therapy With or Without Home Based Intensive Bimanual Training on Clinical Outcomes in Cerebral Palsy Children

DETAILED DESCRIPTION:
Cerebral Palsy is one of the most common issue seen in pediatric rehabilitation .Home based intensive Bimanual training has proven to be one of the most effective rehabilitation training for improving motor. The study determines the effectiveness of routine physical therapy with or without home-based intensive bimanual training on coordination of hands and daily activities of daily living. A nine months randomized control trial was comprised of thirty children with unilateral spastic cerebral palsy aged between 4 to 7 years. One group received routine physical therapy and the other group received a goal specific bimanual training from their parents in their home setting for 3.5 hours per week for 6 weeks according to a modified set up. Follow up sessions were done at 6th week. Activities of daily living and coordination were measured using Pediatric motor log activity scale and ABILHAND respectively.

ELIGIBILITY:
Inclusion Criteria:

* Spastic CP children

  * Both male and female
  * Age 4-7 years
  * Actively grasp of objects from table i.e., stuff toys, making blocks
  * One to one attention

Exclusion Criteria:

* Cognitive delays preventing the child from following two-step instructions

  * Health diagnoses unassociated with USCP.
  * Parents unable to commit to entire duration of intervention.
  * Visual difficulties preventing performance of intervention tasks.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2020-03-06 (Actual); Primary Completion 2020-12-06 (Actual); Study Completion 2020-12-06 (Actual)

PRIMARY OUTCOMES:
ABILHAND | 6th week
  hand coordination

SECONDARY OUTCOMES:
Pediatric Motor Log Activity Scale | 6th week
  Activity of Daily Living

CONTACTS AND LOCATIONS:
Overall Officials: Fatima Ejaz, MS-PT, Principal Investigator — University of Lahore
Locations (1):
- University of lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Results of the study

REFERENCES:
- [Background] Oskoui M, Coutinho F, Dykeman J, Jette N, Pringsheim T. An update on the prevalence of cerebral palsy: a systematic review and meta-analysis. Dev Med Child Neurol. 2013 Jun;55(6):509-19. doi: 10.1111/dmcn.12080. Epub 2013 Jan 24. PMID 23346889
- [Background] Tronnes H, Wilcox AJ, Lie RT, Markestad T, Moster D. Risk of cerebral palsy in relation to pregnancy disorders and preterm birth: a national cohort study. Dev Med Child Neurol. 2014 Aug;56(8):779-85. doi: 10.1111/dmcn.12430. Epub 2014 Mar 13. PMID 24621110
- [Result] Patel DR, Neelakantan M, Pandher K, Merrick J. Cerebral palsy in children: a clinical overview. Transl Pediatr. 2020 Feb;9(Suppl 1):S125-S135. doi: 10.21037/tp.2020.01.01. PMID 32206590
- [Result] He P, Chen G, Wang Z, Guo C, Zheng X. Children with motor impairment related to cerebral palsy: Prevalence, severity and concurrent impairments in China. J Paediatr Child Health. 2017 May;53(5):480-484. doi: 10.1111/jpc.13444. Epub 2017 Jan 17. PMID 28094881